CLINICAL TRIAL: NCT05513924
Title: Efficacy of Topical 5-fluorouracil Versus Topical Latanoprost With Microneedling in Localized Stable Vitiligo: A Randomised Clinical Trial
Brief Title: Comparative Study Between Topical 5-fluorouracil and Latanoprost in Vitiligo.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Amal Mohamed Abdelaziz Ashour, Principal Investigator, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 370
Record Dates: First submitted 2022-08-20; First posted 2022-08-24 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo | interventions — Latanoprost; Ophthalmic Solutions; Fluorouracil

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (topical latanoprost) (Active Comparator): 20 vitiligo patients will receive topical latanoprost solution (the concentration of the solution is 0.005%, pharmaceutically available eye-drop formulation)
  Interventions: Drug: Latanoprost 0.005% Ophthalmic Solution
- Group B (topical 5-fluorouracil) (Active Comparator): 20 vitiligo patients will receive topical 5-fluorouracil 5% solution available as ampoules (Utoral®, EIMC United Pharmaceuticals, Egypt)
  Interventions: Drug: 5Fluorouracil

INTERVENTIONS:
Drug: Latanoprost 0.005% Ophthalmic Solution — The affected area cleaned with betadine surgical solution followed by alcohol 70%.
  Local anesthetic, pridocaine cream, applied on the treated area under occlusion for 30 min before the procedure.
  Using automated microneedling device (Dr Pen Derma Pen Ultima A6®) , which has a disposable head that personalized for each patient and sterilized after each session.
  The derma pen will penetrate the skin with variable depths ranging from 0.25 to 0.5 mm (not more than the depth of the epidermis). It will pass vertically over the vitiligo area in a circular pattern until pinpoint bleeding appears.
  The LT solution will be applied immediately to vitiligo patch one drop (contains 1.5 μg of LT) for every 2.5 cm.
  This procedure will be repeated every two weeks for six months.
  Other Names: Microneedling using Dr Pen Derma Pen Ultima A6®
  Arms: Group A (topical latanoprost)
Drug: 5Fluorouracil — The affected area cleaned with betadine surgical solution followed by alcohol 70%.
  Local anesthetic, pridocaine cream, applied on the treated area under occlusion for 30 min before the procedure.
  Using automated microneedling device (Dr Pen Derma Pen Ultima A6®) , which has a disposable head that personalized for each patient and sterilized after each session.
  The derma pen will penetrate the skin with variable depths ranging from 0.25 to 0.5 mm (not more than the depth of the epidermis). It will pass vertically over the vitiligo area in a circular pattern until pinpoint bleeding appears.
  Topical application of 5-fluorouracil 5% solution will be rubbed over the affected area for about 2 minutes. Occlusive dressing for hours.
  This procedure will be repeated every two weeks for six months.
  Other Names: Microneedling using Dr Pen Derma Pen Ultima A6®
  Arms: Group B (topical 5-fluorouracil)

SUMMARY:
This study aims to compare the efficacy of topical 5-fluorouracil versus topical latanoprost after skin microneedling in the induction of skin repigmentation in localized stable vitiligo patients.

DETAILED DESCRIPTION:
Vitiligo is an acquired pigmentary disorder characterized by depigmented macules and patches secondary to the loss of functional melanocytes. It is a chronic disease that affects between 0.1% and 2% of the general population, affecting both sexes and all races.

Theories regarding loss of melanocytes are based on autoimmune, cytotoxic, oxidant-antioxidant and neural mechanisms.

Therapeutic strategies for vitiligo include nonsurgical and surgical methods. Nonsurgical options include topical corticosteroids and topical calcineurin inhibitors. Phototherapy as psoralen and ultraviolet A (PUVA) and narrow-band ultraviolet B (NB-UVB).

Two types of surgical techniques are available: tissue grafts and cellular grafts, within between autologous cultured epithelial grafts.

Microneedling is a method of transdermal drug delivery using a microneedling device applied to the skin for creating transport pathways through the stratum corneum, increasing the absorption of drugs and decreasing the duration of therapy. In addition, microneedling keeps the epidermis partially intact, fastens recovery, and limits the risk of infection and scarring. 5-Fluorouracil (5-FU) is a chemotherapeutic agent used in the treatment of many malignant tumors and it has been approved for topical use in the treatment of several dermatologic disorders. Localized hyperpigmentation occurred as a side effect of 5-FU use in cancer treatment attracts the attention toward its application in inducing repigmentation in vitiligo patches.

Latanoprost (LT), a prostaglandin F2 alpha analogue used in the treatment of glaucoma, was found to induce skin pigmentation in guinea pigs in addition to its known periocular and iridal pigmentation side effect.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes with stable localized vitiligo : patches should not have any increase or decrease in size or pigmentation for at least 3 months.

Exclusion Criteria:

* Pregnant or lactating female.
* Active Koebner's phenomenon.
* Age less than 10 years.
* All patients included had not received any local or systemic medication for at least 2 months before the study.
* Keloidal tendency.

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Assessment of clinical repigmentation changes of vitiligo lesions according to Physician's Global Assessment [PGA] | 6 months
  5 scales are : G4 (excellent: >75% repigmentation) G3 (very good: 50%-75% repigmentation) G2 (good: 25%-50%) G1 (satisfactory: <25% repigmentation) G0 (poor: no repigmentation)

CONTACTS AND LOCATIONS:
Overall Officials: Hassan M Ibrahim, professor, Study Chair — South Valley University
Locations (1):
- South Valley University, Qina, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bacigalupi RM, Postolova A, Davis RS. Evidence-based, non-surgical treatments for vitiligo: a review. Am J Clin Dermatol. 2012 Aug 1;13(4):217-37. doi: 10.2165/11630540-000000000-00000. PMID 22423621
- [Background] Laddha NC, Dwivedi M, Mansuri MS, Gani AR, Ansarullah M, Ramachandran AV, Dalai S, Begum R. Vitiligo: interplay between oxidative stress and immune system. Exp Dermatol. 2013 Apr;22(4):245-50. doi: 10.1111/exd.12103. Epub 2013 Feb 21. PMID 23425123
- [Background] van Geel N, Ongenae K, Naeyaert JM. Surgical techniques for vitiligo: a review. Dermatology. 2001;202(2):162-6. doi: 10.1159/000051626. PMID 11306848
- [Background] Prausnitz MR. Microneedles for transdermal drug delivery. Adv Drug Deliv Rev. 2004 Mar 27;56(5):581-7. doi: 10.1016/j.addr.2003.10.023. PMID 15019747
- [Background] Prince GT, Cameron MC, Fathi R, Alkousakis T. Topical 5-fluorouracil in dermatologic disease. Int J Dermatol. 2018 Oct;57(10):1259-1264. doi: 10.1111/ijd.14106. Epub 2018 Jun 25. PMID 30187924
- [Background] Mohamed HA, Mohammed GF, Gomaa AH, Eyada MM. Carbon dioxide laser plus topical 5-fluorouracil: a new combination therapeutic modality for acral vitiligo. J Cosmet Laser Ther. 2015;17(4):216-23. doi: 10.3109/14764172.2014.1003241. Epub 2015 Jan 30. PMID 25549816
- [Background] Anbar TS, El-Ammawi TS, Abdel-Rahman AT, Hanna MR. The effect of latanoprost on vitiligo: a preliminary comparative study. Int J Dermatol. 2015;54(5):587-93. doi: 10.1111/ijd.12631. Epub 2014 Dec 29. PMID 25545321
- [Background] Nugroho H, Fadzil MH, Yap VV, Norashikin S, Suraiya HH. Determination of skin repigmentation progression. Annu Int Conf IEEE Eng Med Biol Soc. 2007;2007:3442-5. doi: 10.1109/IEMBS.2007.4353071. PMID 18002737